CLINICAL TRIAL: NCT01755325
Title: Phase III Study of Compound Realgar Formula Realgar-Indigo Naturalis Plus Imatinib Versus Placebo Plus Imatinib in Adult Patients With Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: Phase III Study of Compound Formula Realgar-Indigo Naturalis Plus Imatinib Versus Placebo Plus Imatinib in Adult CML-CP Patients With Ph+
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: not enough patients
Sponsor: Junmin Li (Other)
Responsible Party: Sponsor-Investigator, Junmin Li, Director of hematology department, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RJ-CYP001
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compound realgar natural indigo Tablet (Experimental): Compound realgar natural indigo Tablet, 65mg/kg/d, from day1 to day14,every 4 weeks.
  imatinib,0.4g,qd
  Interventions: Drug: Compound realgar natural indigo Tablet
- placebo (Placebo Comparator): placebo tablet,65mg/kg/d, from day1 to day14,every 4 weeks.
  imatinib 0.4g qd
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Compound realgar natural indigo Tablet — Compound realgar natural indigo Tablet, 65mg/kg/d, from day1 to day14,every 4 weeks.
  imatinib,0.4g,qd
  Arms: Compound realgar natural indigo Tablet
Drug: placebo
  Arms: placebo

SUMMARY:
It is an open-label, randomized, double blind, placebo-controlled parallel-group, multi-center study to evaluate the efficacy and safety of Compound realgar formula Realgar-Indigo naturalis Tablet combined with Imatinib will be compared with imatinib alone in adult patients with diagnosed Philadelphia chromosome-positive (Ph+) chronic myelogenous leukemia in the chronic phase (CML-CP).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age >= 18 years and <= 75 years.
2. Eastern Cooperative Oncology Group （ECOG） performance status (PS) score 0, 1, or 2.
3. Diagnosis of chronic myelogenous leukemia in chronic phase with confirmation of Philadelphia chromosome positive.(Ph+ CML-CP)
4. Ph+ Chronic myelogenous leukemia in chronic phase patients within the first 12 months of diagnosis.
5. Adequate end organ function as defined by:

(1). Alanine transaminase（ALT）, Aspartate transaminase（AST） <=2.5 x upper limit of normal（ULN）.

(2). Total bilirubin <= 1.5 x ULN. (3).Cr <= 1.5 x ULN. (4). Serum amylase and lipase <= 1.5 x ULN. 6. Signed informed consent.

Exclusion Criteria:

1. Previously received or be receiving any of the following medical treatment for CML:

1. . Treatment with Busulfan within 1 day prior to study entry.
2. . Treatment with interferon-alpha within 2 days prior to study entry.
3. . Treatment with hydroxyurea within 1 day prior to study entry.
4. . Treatment with homoharringtonine within 14 days prior to study entry.
5. . Treatment with Cytosine arabinoside within 28 days prior to study entry.
6. . Surgery (Including hematopoietic stem cell transplantation therapy)
7. . Treatment with anthracyclines, or etoposide within 21 days prior to study entry.

2. Treatment with any tyrosine kinase inhibitor(s) or arsenic reagent prior to study entry 3. Patients who are: (a) pregnant, (b) breast feeding, (c) female or male of childbearing potential unwilling to use contraceptive precautions throughout the trial.

4. Major surgery within 4 weeks prior to randomization or who have not recovered from prior surgery.

5. Patients who have not recovered from toxic reaction of prior similar treatment evaluated by investigators.

6. Impaired cardiac function including any one of the following:

1. LVEF < 45%.
2. . Complete left bundle branch block.
3. . Use of a ventricular-paced pacemaker.
4. . Congenital long QT syndrome.
5. . History or presence of ventricular, clinically significant atrial tachyarrhythmias
6. . History or presence of clinically significant bradyarrhythmia.(heart rate persistently less than 50/min)
7. . QTcF > 450 msec for male or 470 msec for female.
8. . History of clinically documented myocardial infarction or unstable angina (during the last 12 month).
9. .Any other severe heart disease. 7. Patients with active, uncontrolled psychiatric disorders, without insight and the ability of exact expression.

8. Uncontrolled medical conditions:

1. .Uncontrolled diabetes with fasting blood-glucose >200mg/dl (11.1mmol/L),or with combined symptoms (nephropathy, peripheral neuropathy).
2. . Uncontrolled hypertension.
3. . Active or uncontrolled infection (persistent fever and worsening of the clinical symptoms) 9. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the tested drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery).

10. History of chronic pancreatitis or history of acute pancreatitis within 1 year of study entry.

11. Acute or chronic uncontrolled liver disease or severe renal disease considered unrelated to CML.

12. Patients actively receiving therapy with strong CYP3A4 inhibitors, strong CYP3A4 inducers or any medications being potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.

13. Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 4 weeks prior to randomization.

14. Known to be allergic to the study drugs, including crude drug or adjuvant. 15. As investigators evaluate, the patients do not fit to join the study (such as with severe complications) .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2012-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of Major molecular response（MMR） at 12 months | 12 months of follow-up from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Saijuan Chen, M.D., Study Chair — Runjin Hospital
Locations (13):
- China (13):
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - The NO.1 People's Hospital of Huaian, Huaian, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - First Hospital Affiliated to Suzhou University, Suzhou, Jiangsu
  - The FIrst Affiliated Hospital, College of Medicine, Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital, College of Medicine, Nanchang University, Nanchang, Jiangxi
  - The Tumor Hospital of Jiangxi, Nanchang, Jiangxi
  - The NO.1 Hospital of Nanchang, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Xijing Hospital-Fourth Military Medical University, Xi'an, Shan'xi
  - The FIrst Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The People's Hospital of Peking University, Beijing
  - Ruijin Hospital, Shanghai